CLINICAL TRIAL: NCT04958850
Title: The Third Epidemiological Research of Refractory Wounds in China
Status: Completed | Type: Observational
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Other Study IDs: 2018-051
Record Dates: First submitted 2021-07-06; First posted 2021-07-12 (Actual); Last update posted 2021-07-12 (Actual); Status verified 2017-11

CONDITIONS: Wound of Skin
Keywords: cutaneous wounds; epidemiology; China

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: a cross-sectional survey — Collect the data of this year and compare it with that of ten years ago

SUMMARY:
This study is a cross-sectional survey in patients who underwent treatment of chronic cutaneous wounds from a nationally representative sample in our hospital from January 2018 to December 2018．

DETAILED DESCRIPTION:
Chronic cutaneous wounds represent a major health care burden in China However, limited information exists regarding the epidemiologic changes associated with recent social and economic devdopment．We designed a cross-sectional survey in patients who underwent treatment of chronic cutaneous wounds from a nationally representative sample in our hospital from January 2018 to December 2018．

ELIGIBILITY:
Inclusion Criteria:

- Patients who underwent treatment of chronic cutaneous wounds in our hospital from 1/2018-12/2018．

Exclusion Criteria:

- No

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Chinese Patients who underwent treatment of chronic cutaneous wounds in our hospital from 1/2018-12/2018
Sampling Method: Probability Sample
Enrollment: 500 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
the prevalence of chronic cutaneous wounds among hospitalized patients | 1 year
  All the patients with refractory wounds on the body surface

SECONDARY OUTCOMES:
cause of disease | 1 year
  diabetes, trauma or other.
Bacterial etiology | 1 year
  patients had results of bacterial cultivation
Treatment expense | 1 year
  Treatment was paid by the patients, social medical insurance, commercial medical insurance, or free medical care．

CONTACTS AND LOCATIONS:
Overall Officials: Han Chunmao, Pro, Study Chair — 2nd Affiliated Hospital, School of Medicine, Zhejiang University
Locations (1):
- 2nd Affiliated Hospital, School of Medicine, Zhejiang University, Hanzhou, Zhejiang, China